CLINICAL TRIAL: NCT06760247
Title: Frequency And Level Of Dental Injury Related To Conventional Direct Laryngoscopy: A Prospective Observational Study
Brief Title: Dental Injury Related To Conventional Direct Laryngoscopy
Acronym: dentalinjury
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, FUNDA ARUN, Asst. Prof., Selcuk University
Other Study IDs: F004
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Asa I-III Patients; Intubated Patients; Laryngoscopy
Keywords: dental trauma; general anesthesia; endotracheal intubation; laryngoscopy
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intubated: intubated by direkt laryngoscopy under general anesthesia
  Interventions: Procedure: intubated general anesthesia with propofol IV, rocuronium IV ,sevoflurane and N2O gas

INTERVENTIONS:
Procedure: intubated general anesthesia with propofol IV, rocuronium IV ,sevoflurane and N2O gas — endotracheal intubation by using direct laryngoscopy
  Other Names: endotracheal intubation

SUMMARY:
This research explores the occurrence of minor dental injuries and their associated effects by employing the transillumination technique with a cold light source. Unlike traditional methods primarily concentrating on major traumas detectable through standard laryngoscopy, this study aims to shed light on the subtler yet potentially impactful dental traumas that may otherwise go unnoticed. Through this innovative approach, investigators hope to gain deeper insights into the nuances of dental damage and its implications for oral health.

DETAILED DESCRIPTION:
This study aims to investigate especially minor dental traumas and associated damages instead of major traumas that can be directly seen due to conventional laryngoscopy using transillumination technique with cold light source.

After the approval of the Selcuk University Local Institutional Ethics Committee (2017/05), 300 ASA I-III adult patients who underwent elective surgical operations under general anesthesia and underwent endotracheal intubation were included in this prospective, double-blinded study. Written informed consent was obtained from each patient during the preoperative anesthetic evaluation.

During the preoperative anesthetic evaluation, an anesthetist and dentist in the study team performed a detailed oral physical examination on all study patients. Demographic data such as age, gender, body weight, height, data related to airway management such as mallampati score, thromental distance, mouth opening size, and information about past anesthesia history, including previously described difficult intubation and medical condition, were questioned, and recorded. During a dental examination, all teeth, but particularly anterior 6 of maxillary and mandibular teeth, were examined regarding general dental hygiene and the existence of any missing teeth, tooth decay, plaque and stone formation, discoloration, gum problems such as recession and gingivitis, and tooth trauma. The patients with the presence of deformation due to a trauma or a congenital abnormality in the maxilla-fascial region, a swinging tooth, and a history of previous surgical operation regarding the maxilla-fascial region and oral cavity were not included in the study.

All patients were subjected to the same anesthetic process. None of the patients were given anesthetic premedication on the day of surgery. Anesthesia induction was achieved with 2.0 mg.kg-1 iv propofol, 2.0 mg.kg-1 iv fentanyl, and 0.6 mg.kg-1 iv rocuronium after routine monitoring with ECG, non-invasive blood pressure, and SpO2. Each patient was ventilated with a face mask with 100% O2 for 2-3 minutes and intubated with a proper endotracheal tube by the same anesthetist using a conventional laryngoscope. All intubations were achieved by anesthesiologists with different statuses (senior assistants and consultants who were blind to the study). After the endotracheal intubation, the anesthesiologist included in the study recorded the data about intubation and airway management such as Cormack-Lehane Score, laryngoscope blade type and size, difficulty in intubation, use of additional devices such as oral airway, intubating supraglottic airway device, video laryngoscope, and intubating guide in the airway management, and the number of intubating attempts by asking the practitioner.

The intraoperative dental evaluation was performed using a transillumination technique with a cold light source at two different time points: T1: Before anesthesia induction, and T2: After endotracheal intubation, before the start of the surgical operation. The same dentist performed all dental evaluations. Although all teeth were evaluated, the evaluation with the cold light source was particularly for every six teeth in the lower and upper jaws.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II,III
* Intubated by direct laringscopy

Exclusion Criteria:

* deformation due to a trauma or a congenital abnormality in the maxilla-fascial region
* a swinging tooth
* history of previous surgical operations regarding the maxilla-fascial region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I_III patients intubated by direct laryngoscopy under general anesthesia
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
dental injury | 1 year
  frequency of dental injury due to direct laryngoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Funda Arun, Asst. Prof., Principal Investigator — Selcuk University
Locations (1):
- Selcuk University Faculty of Dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to private conditions, we do not plan to share IPD with other researchers. This decision is based on data confidentiality, participant privacy, and compliance with ethical and regulatory guidelines. While IPD sharing is not part of our plan, we are open to providing aggregate data or summary results if you'd like to.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT06760247/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT06760247/ICF_001.pdf